CLINICAL TRIAL: NCT01809054
Title: Pilot Study Evaluating Alterations in Thrombogenicity and Platelet Reactivity Following Lower Extremity Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LifeBridge Health (Other)
Collaborators: Haemonetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1888
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Primary Total Hip and Knee Arthroplasty
Keywords: Hip, Knee, Arthroplasty, venous thromboembolic events, blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Fondaparinux; Intermittent Pneumatic Compression Devices; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arixtra Arm (Active Comparator): Arixtra (2.5 mg SQ/QD) subcutaneous injection daily for 2 weeks followed by aspirin 325 mg for 5 weeks
  Interventions: Drug: Arixtra; Drug: Aspirin
- Pneumatic compression stockings arm (Active Comparator): Pneumatic compression stockings (MCS, Active Care, medical compression systems Inc., Israel) for 2 weeks with concomitant Aspirin 325 mg daily for 5 weeks.
  Interventions: Device: Pneumatic compression stockings; Drug: Aspirin

INTERVENTIONS:
Drug: Arixtra
  Arms: Arixtra Arm
Device: Pneumatic compression stockings — Pneumatic compression stockings (MCS, Active Care, medical compression systems Inc., Israel)
  Arms: Pneumatic compression stockings arm
Drug: Aspirin

SUMMARY:
This is a prospective, randomized study from pre-surgery to 6 weeks post-surgery designed to detect changes in coagulability following elective total knee and hip arthroplasty. Patients will be randomized to one of the two standard prophylaxis treatments used at Sinai Hospital:

1. Arixtra (2.5 mg SQ/QD) subcutaneous injection daily for 2 weeks followed by aspirin 325 mg for 5 weeks, or
2. Pneumatic compression stockings (MCS, Active Care, medical compression systems Inc., Israel) for 2 weeks with concomitant Aspirin 325 mg daily for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women age ≥ 18 years old
2. Total knee or total hip arthroplasty planned in the 60 days following study enrollment

Exclusion Criteria:

1. Pre-existing anti-coagulant therapy (Heparin, Lovenox, Arixtra, Warfarin, Xarelto, and all other non-mentioned anticoagulants) on admission
2. History of bleeding diathesis
3. Known active malignancy
4. Prothrombin time >1.5 x control
5. Platelet count < 100,000/mm3, hematocrit < 30%, creatinine clearance <30 mL/min
6. Immunosuppression, e.g., human immunodeficiency virus (HIV) infection, Chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, Bacterial endocarditis
7. Major surgery within past 3 months of enrollment
8. Patients requiring bilateral arthroplasty
9. Body weight <50 kg (venous thromboembolism prophylaxis only)
10. Unable to return to site for follow-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rubin Institute for Advanced Orthopedics, Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sinai Center for Thrombosis Research, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Arixtra Arm: Arixtra (2.5 mg SQ/QD) subcutaneous injection daily for 2 weeks followed by aspirin 325 mg for 5 weeks
  Arixtra
  Aspirin
- Pneumatic Compression Stockings Arm: Pneumatic compression stockings (MCS, Active Care, medical compression systems Inc., Israel) for 2 weeks with concomitant Aspirin 325 mg daily for 5 weeks.
  Pneumatic compression stockings: Pneumatic compression stockings (MCS, Active Care, medical compression systems Inc., Israel)
  Aspirin
Period: Overall Study
Arm/Group | Arixtra Arm | Pneumatic Compression Stockings Arm
Started | 27 | 22
Completed | 27 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arixtra Arm | Pneumatic Compression Stockings Arm | Total
Number analyzed (Participants) | 27 | 22 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13) | 58 (14) | 58 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Blood Loss
Description: requiring transfusion
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Arixtra Arm | Pneumatic Compression Stockings Arm
Number analyzed (Participants) | 27 | 22
participants | 6 | 1

2. Secondary Outcome: Deep Vein Thrombosis
Description: verified by ultrasound
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Arixtra Arm | Pneumatic Compression Stockings Arm
Number analyzed (Participants) | 27 | 22
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arixtra Arm | Pneumatic Compression Stockings Arm
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes